CLINICAL TRIAL: NCT01525992
Title: A Community Pharmacy-based Intervention on Type 2 Diabetic Patients to Improve Medications Adherence and Disease Outcomes; a Randomized Controlled Trial.
Brief Title: A Community Pharmacy-based Program to Improve Management of Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Research Center for Rational Use of Drugs (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 90-04-156-16161
Record Dates: First submitted 2012-01-31; First posted 2012-02-03 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Community Pharmacy Services; Pharmacists; Diabetes Mellitus; Diabetes Mellitus, Type 2; Self Care; Randomized Controlled Trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Community Pharmacy-based Program (Experimental)
  Interventions: Behavioral: Community pharmacist-led diabetes education program
- Usual care (Active Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Community pharmacist-led diabetes education program — A trained pharmacist will counsel each patient based on his/her individual needs about medications, life style and self-care. The pharmacist will use a checklist to document the type of education delivered to each patient. A glucometer is provided for each patient in this arm to monitor blood glucose daily. Three to six visits to the community pharmacy are set during the 6-months study period. At each visit, medication related problems and self-care issues are discussed with the patient and the glucometer test strips are provided for the following month. A telephone call will be made to each patient between visits to ensure adherence to drug therapy and resolve any problems .
  Arms: Community Pharmacy-based Program
Other: Usual care — The baseline and 6-month follow-up visits to the community pharmacy will be required. If the physician prefers more visits to his office during the study period, it will be granted. The glucometer and a training session about diabetes self-care will be provide at the end of study for control group patients.
  Arms: Usual care

SUMMARY:
In this study the investigators aim to evaluate the impact of a community pharmacy-based program to educate type 2 diabetic patients about medications, life style and self-care.

DETAILED DESCRIPTION:
Diabetes mellitus type 2 is a progressive metabolic disorder that leads to several morbidities and increased mortality and costs. Studies showed that strict control of blood glucose in diabetic patients reduces patients' risk of microvascular complications. Community pharmacies are a well-placed healthcare facility located at the heart of the community with convenient access to pharmacists as health care professionals. Some studies have shown effective interventions led by community and clinical pharmacist in developed countries. In developing countries, little evidence exists about feasibility of implementing community pharmacy-based services to promote medications adherence, self glucose monitoring and self-care in diabetic patients.

This study is a 2 arm randomized controlled trial. Eligible patients are referred to the community pharmacy from an endocrinologist's office. Of 135 type-2 diabetic patients who will be recruited in the study,68 will be randomly allocated to the intervention arm using telephone balanced blocked randomization method.

A community pharmacy-based program will provide training about medications, life style and self-care to the intervention arm. The control arm (67 patients) will receive usual care during the study period.

The primary outcome of this study is measured as change in hemoglobin A1C pre and post intervention. As the secondary outcome, medications adherence, diabetes self-care activity, body mass index and blood pressure are measured.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients using oral anti diabetic medications.
* Hemoglobin A1c > 7 within the previous month before recruitment
* Adequate literacy and ability to use the glucometer.
* Signing the informed consent

Exclusion Criteria:

* Patients requiring adjunct insulin therapy.
* Patients with concurrent heart failure (stage 4).
* Patients who fast in Ramadan.
* Patients receiving diabetes education in other programs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-03; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | Change from baseline (at the point of recruiting) Hemoglobin A1c at 6 months.
  Hemoglobin A1c is measured in all patients prior to participating in the study. All patients will be required to take the test again at the end of the study (6 months) .

SECONDARY OUTCOMES:
Medication adherence | Change from baseline (at the point of recruiting) medication adherence at 6 months.
  Medication adherence will be measured using "Morisky Medication Adherence Questionnaire" which will be translated into Farsi.The validity and reliability of the translated questionnaire will be investigated primarily.
Self-care activity | Change from baseline (at the point of recruiting) Self-care activity at 6 months.
  Self-care activity will be measured using "Diabetes Self-care Activity Measure" questionnaire which will be translated into Farsi. We will investigate the validity and reliability of the translated questionnaire.
Body Mass Index | Change from baseline (at the point of recruiting) Body Mass Index at 6 months.
  Weight (measured in kilograms) divided by square of height (measured in Meters).
Blood pressure | Change from baseline (at the point of recruiting) Blood pressure at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Kheirollah Gholami, M.Sc, PharmD, Study Chair — Tehran University of Medical Sciences; Zahra Jahangard-Rafsanjani, PharmD, Study Director — Tehran University of Medical Sciences; Arash Rashidian, MD, Ph.D, Principal Investigator — Tehran University of Medical Sciences; Navid Saadat, MD, Principal Investigator — Shahid Beheshti University of Medical Sciences; Amir Sarayani, PharmD, MPH, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Taleghani Community Pharmacy, Faculty of Pharmacy, Tehran University of Medical Sciences, Tehran, Tehran Province, Iran